CLINICAL TRIAL: NCT02943135
Title: Effect of Self-administered Lidocaine In-situ Gel on Intrauterine Device Insertion Pain: A Randomized Controlled Trial
Brief Title: Lidocaine In-situ Gel Before Intrauterine Device Insertion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LISID
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pain Relief

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine in-situ (Active Comparator): Self-administered gel 10 min before intrauterine device insertion
  Interventions: Drug: lidocaine in-situ gel
- placebo (Placebo Comparator): Self-administered gel 10 min before intrauterine device insertion
  Interventions: Drug: placebo in-situ gel

INTERVENTIONS:
Drug: lidocaine in-situ gel — lidocaine in-situ gel
  Arms: lidocaine in-situ
Drug: placebo in-situ gel — placebo in-situ gel
  Arms: placebo

SUMMARY:
Intrauterine device can cause pain and discomfort in several ways: Use of the tenaculum to grasp the cervix and straighten the uterus for proper insertion; trans-cervical actions including measuring uterine depth, inserting the insertion tube, and removing the tube; and placement of the device in the uterus.

ELIGIBILITY:
Inclusion Criteria:

* Women not taken analgesics or anxiolytics in the 24 hours prior insertion
* Women not taken misoprostol prior to insertion
* No contraindication to or history of allergic reaction to lidocaine
* Women who will accept to participate in the study

Exclusion Criteria:

* Lidocaine allergy
* Any contraindication to device placement

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Mean pain score during intrauterine device insertion | 30 min

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Ahmed Abbas, Assiut, Cairo Governorate
  - Assiut University, Asyut

IPD SHARING:
Plan to Share IPD: Undecided